CLINICAL TRIAL: NCT02646345
Title: WHO Surgical Safety Checklist Implementation and Its Impact in Perioperative Morbidity and Mortality in an Academic Medical Center in Chile
Brief Title: Surgical Checklist Success in Latin America
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 12-218
Record Dates: First submitted 2015-12-28; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: External Causes of Morbidity and Mortality; External Causes of Morbidity (V00-Y99)
Keywords: Checklist; Mortality; Latin America; Surgery; Morbidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre Checklist: All surgical encounters before surgical checklist implementation
- Post Checklist: All surgical encounters after surgical checklist implementation
  Interventions: Procedure: Surgical checklist

INTERVENTIONS:
Procedure: Surgical checklist — Use of the World Health Organization Surgical checklist
  Groups: Post Checklist

SUMMARY:
Limited information is available about surgical checklist effectiveness in Latin America. We plan to compare the pre and post surgical checklist implementation in a tertiary healthcare center in terms of morbidity (length of stay and surgical site infection rate) and in-hospital mortality rate.

DETAILED DESCRIPTION:
The purpose was to determine the impact of the implementation of the World Health Organization (WHO) Surgical Safety Checklist in terms of morbidity and mortality in adult surgical patients in a tertiary healthcare institution in Chile.

After Institutional Review Board (IRB) approval (Facultad de Medicina, Pontificia Universidad Católica de Chile, Santiago, Chile), a retrospective analysis of all surgical encounters on patients age 15 and above from January 2005 to December 2012 at our center will be reviewed.

Encounter data will include up to 14 diagnostic and procedure International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) codes, demographic data, date of admission and discharge, emergency status, healthcare system used and in-hospital death. A 5-level "high risk" variable was created in order to account for surgical complexity and associated in-hospital mortality (level 1, surgeries with <1% in-hospital mortality; level 2, 1% to <5%; level 3, 5% to <10%; level 4, 10% to <15%; level 5, > or = 15%)6.

Surgical heterogeneity will be calculated by the Internal Herfindahl Index, which represents the diversity or comprehensiveness of the types of procedures performed at a facility.

Statistics:

Propensity score (PS) analysis will be used to control for differences in baseline characteristics. The PS is the conditional probability of receiving an exposure (e.g. checklist) given a set of measured covariates. To estimate the PS, a logistic regression model will be used in which "treatment" status (checklist performed vs. not performed) will be regressed on the baseline (pre-treatment) characteristics.

PS analysis will be implemented in two ways to control for confounding:

1. PS matching: matching will be performed using a one-to-one nearest neighbor caliper matching without replacement with a caliper size of 0.2 standard deviations. Balances in the distribution of baseline covariates will be assessed by estimating absolute standardized differences of the covariates between the two groups before and after matching. Any imbalanced covariates (standardized difference >10%) after matching will be adjusted for in the final analysis. As the PS matched sample does not consist of independent observations, we will use a marginal regression model with robust standard errors.
2. PS weighting: the entire sample will be weighted by the inverse probability of the treatment weights derived from the PS. If a subject has a higher probability of being in a group, it will be considered over-represented and therefore will be assigned a lower weight. Conversely, if the subject has a smaller probability, it will be considered as under-represented and will be assigned a higher weight. We then will fit a weighted linear regression model using an indicator variable representing checklist intervention status as the sole predictor, and mortality as our outcome variable.

Data will be expressed as mean (SD; standard deviation) or median (IQR, interquartile range) unless otherwise stated. A two-sided p value less than 0.05 will be considered significant. The analyses will be performed using STATA v.12.0 (StataCorp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* All surgical patients

Exclusion Criteria:

* Obstetrical patients delivering vaginally
* Patients less than 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All surgical patients age 15 and above
Sampling Method: Probability Sample
Enrollment: 70639 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mortality | Three years
  30 day postoperative mortality

SECONDARY OUTCOMES:
Morbidity | Three years
  30 day postoperative surgical site infection (measured in number of patients with surgical site infection)
Length of stay | Three years
  Length of stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Hector J Lacassie, MD, Principal Investigator — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] de Vries EN, Ramrattan MA, Smorenburg SM, Gouma DJ, Boermeester MA. The incidence and nature of in-hospital adverse events: a systematic review. Qual Saf Health Care. 2008 Jun;17(3):216-23. doi: 10.1136/qshc.2007.023622. PMID 18519629
- [Background] Tscholl DW, Weiss M, Kolbe M, Staender S, Seifert B, Landert D, Grande B, Spahn DR, Noethiger CB. An Anesthesia Preinduction Checklist to Improve Information Exchange, Knowledge of Critical Information, Perception of Safety, and Possibly Perception of Teamwork in Anesthesia Teams. Anesth Analg. 2015 Oct;121(4):948-956. doi: 10.1213/ANE.0000000000000671. PMID 25806399
- [Background] Schwarze ML, Barnato AE, Rathouz PJ, Zhao Q, Neuman HB, Winslow ER, Kennedy GD, Hu YY, Dodgion CM, Kwok AC, Greenberg CC. Development of a list of high-risk operations for patients 65 years and older. JAMA Surg. 2015 Apr;150(4):325-31. doi: 10.1001/jamasurg.2014.1819. PMID 25692282
- [Background] Wachtel RE, Dexter F. Differentiating among hospitals performing physiologically complex operative procedures in the elderly. Anesthesiology. 2004 Jun;100(6):1552-61. doi: 10.1097/00000542-200406000-00031. PMID 15166578
- [Background] Urbach DR, Govindarajan A, Saskin R, Wilton AS, Baxter NN. Introduction of surgical safety checklists in Ontario, Canada. N Engl J Med. 2014 Mar 13;370(11):1029-38. doi: 10.1056/NEJMsa1308261. PMID 24620866
- [Background] de Vries EN, Prins HA, Crolla RM, den Outer AJ, van Andel G, van Helden SH, Schlack WS, van Putten MA, Gouma DJ, Dijkgraaf MG, Smorenburg SM, Boermeester MA; SURPASS Collaborative Group. Effect of a comprehensive surgical safety system on patient outcomes. N Engl J Med. 2010 Nov 11;363(20):1928-37. doi: 10.1056/NEJMsa0911535. PMID 21067384
- [Background] Calland JF, Turrentine FE, Guerlain S, Bovbjerg V, Poole GR, Lebeau K, Peugh J, Adams RB. The surgical safety checklist: lessons learned during implementation. Am Surg. 2011 Sep;77(9):1131-7. PMID 21944620
- [Background] Leape LL. The checklist conundrum. N Engl J Med. 2014 Mar 13;370(11):1063-4. doi: 10.1056/NEJMe1315851. No abstract available. PMID 24620871
- [Background] Conley DM, Singer SJ, Edmondson L, Berry WR, Gawande AA. Effective surgical safety checklist implementation. J Am Coll Surg. 2011 May;212(5):873-9. doi: 10.1016/j.jamcollsurg.2011.01.052. Epub 2011 Mar 12. PMID 21398154